CLINICAL TRIAL: NCT07122505
Title: Oromyofunctional Training: an Innovative Rehabilitation Program for Pediatric Obstructive Sleep Apnea
Brief Title: Oromyofunctional Therapy: a Rehabilitation Program for OSA in Children With Down Syndrome and Prader-Willi Syndrome
Acronym: OROFIT-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Organization: University Hospital, Ghent (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2024-0002
Record Dates: First submitted 2025-04-28; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea (OSA); Orofacial Myofunctional Disorders
Keywords: Orofacial myofunctional therapy; Obstructive sleep apnea; Down syndrome; Prader-Willi syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome; Prader-Willi Syndrome | interventions — Myofunctional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OSA-patients (Experimental): orofacial myofunctional therapy
  Interventions: Behavioral: Orofacial myofunctional therapy

INTERVENTIONS:
Behavioral: Orofacial myofunctional therapy — Orofacial myofunctional therapy consists of a set of oropharyngeal exercises to correct abnormal orofacial functions such as mouth breathing and a caudal tongue position, and strengthen upper airway muscles (e.g., muscles of the tongue and soft palate) that are involved in maintaining airway patency.
  Other Names: Oromyofunctional therapy; Oropharyngeal exercises

SUMMARY:
Obstructive sleep apnea (OSA) is a prevalent medical condition with important implications for overall health and quality of life in both children. Therefore, it is important to treat OSA early and effectively. Children with Down syndrome and Prader-Willi syndrome have many predisposing factors for OSA, including mouth breathing, narrow upper airways resulting from craniofacial abnormalities, and generalized hypotonia, which increases UA collapsibility and multilevel obstructions. Adenotonsillectomy is the first-line treatment. Unfortunately, up to 55% of children with Down syndrome and up to 79% of children with Prader-Willi syndrome suffer from residual OSA after adenotonsillectomy. Therefore, exploring other treatment options for these children is an interesting and relevant avenue for research.

This study will evaluate the effectiveness of orofacial myofunctional therapy as a treatment option for children with Down syndrome or Prader-Willi syndrome and obstructive sleep apnea. Orofacial myofunctional therapy consists of a set of oropharyngeal exercises to correct abnormal orofacial functions and strengthen upper airway muscles that are involved in maintaining airway patency. Both objective and subjective/patient-reported outcomes are collected to obtain a comprehensive understanding of the potential of orofacial myofunctional therapy as a treatment for OSA.

DETAILED DESCRIPTION:
Objective: Determine the effect of 20 weeks of orofacial myofunctional therapy on oromyofunctional, sleep and sleep-related quality of life outcomes in children with OSA (AHI > 1) and Down syndrome or Prader-Willi syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4-18
* Diagnosed with Down syndrome or Prader-Willi syndrome
* Diagnosed with Obstructive Sleep Apnea on Polysomnography (AHI<1)

Exclusion criteria:

* History of Orofacial Myofunctional Therapy
* Undergoing an orthodontic procedure during the study period
* Undegoing an OSA treatment during the study period
* Orofacial congenital deformities (not related to Down syndrome or Prader-Willi syndrome)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Sleep: change in OAHI | measurement 1: pre therapy, measurement 2: post therapy (after 20 weeks of therapy)
  Obstructive apnea hypopnea index measured by polysomnography

SECONDARY OUTCOMES:
Orofacial Myofunctional Outcomes: OMES score | measurement 1: pre therapy, measurement 2: post therapy (after 20 weeks of therapy)
  core on the 'Orofacial Myofunctional Evaluation with scores' protocol.
Orofacial strength | measurement 1: pre therapy, measurement 2: post therapy (after 20 weeks of therapy)
  Lip and tongue strength measured with the Iowa Oral Performance Instrument.
Quality of Life outcomes: CHQ-PF28 | measurement 1: pre therapy, measurement 2: post therapy (after 20 weeks of therapy)
  Child Health Questionnaire (CHQ-PF28)
Sleep: PSQ | measurement 1: pre therapy, measurement 2: post therapy (after 20 weeks of therapy)
  Score on the Pediatric Sleep Questionnaire
Sleep: BSQ | measurement 1: pre therapy, measurement 2: post therapy (after 20 weeks of therapy)
  Score on the Berlin Sleep Questionnaire
Sleep: PSG | measurement 1: pre therapy, measurement 2: post therapy (after 20 weeks of therapy)
  Polysomnography: - Oxygen Desaturation Index - Saturation 93% - Minimum saturation - Mean saturation - Sleep efficiency - Apnea Index (AI) (- Apnea-Hyponea Index (AHI) = primary outcome derived from PSG)

CONTACTS AND LOCATIONS:
Overall Officials: Kristiane Van Lierde, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No